CLINICAL TRIAL: NCT04157972
Title: Short-term Effects of SIMEOX on Static Hyperinflation in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of SIMEOX on Static Hyperinflation in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, William Poncin, PT, PhD, Principal Investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SIMEOX-004
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: The visits include sessions (test 1 and 2) with SIMEOX or a positive expiratory pressure device (PEP) (chosen according to the subject's randomization) lasting 20 minutes, each followed by a rest period of 30 minutes.
  Lung function tests will be performed before, after and 30 minutes after performing the devices (SIMEOX and PEP).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIMEOX (Active Comparator): Participants will have to perform 20 minutes of SIMEOX. Passive exhalation is required using the SIMEOX, starting from tidal volume and going until achieving residual volume.
  Interventions: Device: SIMEOX
- PEP (Active Comparator): Participants will have to perform 20 minutes of PEP. Active exhalation is required using a PEP device, starting from tidal volume and going until achieving residual volume.
  Interventions: Device: PEP

INTERVENTIONS:
Device: SIMEOX — SIMEOX is a device generating a succession of gentle depression at the mouth.
  Arms: SIMEOX
Device: PEP — A PEP device (Pari-PEP) will be used to provoke a positive expiratory pressure while exhaling, thereby stabilizing the airways during expiration.
  Arms: PEP

SUMMARY:
This study will investigate the effects on the SIMEOX technology on static hyperinflation in patients with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
This is a crossover study assessing the short-term effects of SIMEOX and PEP device on static hyperinflation in patients with COPD.

Patients will perform lung function tests (to assess the residual volume and functional residual capacity) before, after and 30 minutes after a 20-min long session of SIMEOX or PEP (depending of randomization).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic obstructive pulmonary disease,
* Forced expiratory volume in 1s (FEV1) <80% of predicted value,
* Stable condition (no pulmonary exacerbation for more than 28 days).

Exclusion Criteria:

* Routine use of one of the two treatments - SIMEOX and/or PEP,
* Inability to understand or carry out the instructions,
* Severe cardiac comorbidity, neuromuscular disease,
* Severe scoliosis,
* Patient with a pacemaker.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Change in functional residual capacity (FRC) using body plethysmography | 15 minutes
  FRCpleth before, after and 30 minutes after performing SIMEOX and PEP will be compared.
Change in functional residual capacity (FRC) using helium dilution | 5 minutes
  FRChe before, after and 30 minutes after performing SIMEOX and PEP will be compared.
Change in air trapping | 20 minutes
  FRCpleth - FRChe before, after and 30 minutes after performing SIMEOX and PEP will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Macedo JRFF, Aubriot AS, Reychler G, Penelle M, Gohy S, Poncin W. The intermittent intrapulmonary deflation technique for airway clearance in patients with cystic fibrosis: A randomized trial. Respir Med Res. 2024 Nov;86:101094. doi: 10.1016/j.resmer.2024.101094. Epub 2024 Feb 29. PMID 38843595
- [Derived] Ribeiro Fonseca Franco de Macedo J, Reychler G, Poncin W, Liistro G. Effects of the intermittent intrapulmonary deflation technique on expiratory flow limitation: an in vitro study. J Clin Monit Comput. 2024 Feb;38(1):69-75. doi: 10.1007/s10877-023-01093-3. Epub 2023 Nov 2. PMID 37917211
- [Derived] de Macedo JRFF, Reychler G, Liistro G, Poncin W. Short-Term Effect of Intermittent Intrapulmonary Deflation on Air Trapping in Patients With COPD. Respir Care. 2023 Apr;68(4):478-487. doi: 10.4187/respcare.10398. Epub 2023 Feb 21. PMID 36810360